CLINICAL TRIAL: NCT01614496
Title: Rule-Based Closed Loop System for Type 1 Diabetes Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Other Study IDs: PS09/01255
Record Dates: First submitted 2012-06-07; First posted 2012-06-08 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Algorithms

INTERVENTIONS:
Other: Algorithm for insulin administration

SUMMARY:
The aim of the study is to assess the efficacy and safety of a Rule-based Closed Loop system, using subcutaneous way, for the overnight and prandial glucose control in type 1 diabetic subjects. Ten subjects will be enrolled and they will participate in a cross-over study with a control night, using their usual insulin pump pattern, and with a experimental night, being controlled for the closed loop system. Each night includes the overnight control and prandial control of the breakfast.

The system proposes an insulin dose every 5 minutes according with the value of glucose displayed by the continuous glucose monitoring system.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes
* Insulin pump treatment
* Undetectable C-Peptide

Exclusion Criteria:

* Autonomous system neuropathy

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Time spent with glucose in the target range

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology and Nutrition Department. Corporació Sanitària i Universitària Parc Taulí, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Capel I, Rigla M, Garcia-Saez G, Rodriguez-Herrero A, Pons B, Subias D, Garcia-Garcia F, Gallach M, Aguilar M, Perez-Gandia C, Gomez EJ, Caixas A, Hernando ME. Artificial pancreas using a personalized rule-based controller achieves overnight normoglycemia in patients with type 1 diabetes. Diabetes Technol Ther. 2014 Mar;16(3):172-9. doi: 10.1089/dia.2013.0229. Epub 2013 Oct 23. PMID 24152323